CLINICAL TRIAL: NCT02816333
Title: Korean Registry of Thoracic Endovascular Aortic Repair Timing for Type B Aortic Dissection (K-TEAM Study): A Prospective Multicenter Registry
Status: Withdrawn | Type: Observational
Why Stopped: Due to the withdrawal of Gore Korea Co.Ltd., manufacturer of medical device, it is impossible to supply the medical device(C-TAG).
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 1-2016-0003
Record Dates: First submitted 2016-06-23; First posted 2016-06-28 (Estimated); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Type B Aortic Dissection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Type B aortic dissection: Patients with Type B aortic dissection requiring TEVAR

SUMMARY:
Prospective, single-arm, multi-center registry study A total of 50 subjects with Type B aortic dissection who meet all inclusion and exclusion criteria will be included.

Patients will be treated with TEVAR using conformable TAG endograft (Gore). Patients will be followed clinically for 12 months after the procedure. CT will be performed at 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. a) In case of acute Type B dissection (14 days from first dissection)

   * Maximum aortic diameter >40 mm or
   * Increase in aortic diameter >2 mm from baseline b) In case of subacute (15~90 days) or chronic (90 days ~ 1 year) Type B
   * Maximum aortic diameter >55 mm or
   * Increase in aortic diameter >4 mm from baseline
2. Age 19-80 years.
3. Aorta anatomy appropriate for stent graft therapy,

   1. Proximal landing zone (diameters between 23 and 42 mm) is not aneurysmal, dissected or significantly thrombosed.
   2. Proximal landing zone length >20 mm (length from the left subclavian artery origin to the primary intima tear or length from the left common carotid artery origin to the primary intima tear when the left subclavian artery is embolized and possibly revascularized), as measured from the outer curve of the aorta.
4. Declaration of voluntary participation in the study with signed informed consent form.

Exclusion Criteria:

1. Endorgan ischemia or evidence of malperfusion due to aortic dissection
2. Aortic rupture or impeding rupture due to aortic dissection
3. Renal dysfunction with serum Cr level >2.0 mg/dL
4. Marfan syndrome, Loeys-Diets, Ehlers-Danlos syndrome, or other connective tissue diseases
5. Uncontrolled active infection or active vasculitis.
6. Recent myocardial infarction or cerebrovascular accident within 4 weeks prior to study enrollment.
7. Previous thoracic aorta surgery or stent-graft implantation
8. Planned concomitant surgical procedures (other than left subclavian artery transposition or bypass) or major surgery within 30 days of study enrolment.
9. Women with positive pregnancy test or at child bearing age
10. Life expectancy <1 year due to comorbidity

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Type B aortic dissection requiring thoracic endovascular aortic repair
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-06; Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Major adverse event | 12 months
  A composite of all-cause death, re-intervention, and aortic dilation > 5 mm in maximal aortic diameter

SECONDARY OUTCOMES:
Aortic remodeling | 12 months
  Change in maximal aorta, true lumen, and false lumen dimensions
Aorta-related complications | 12 months
  composite events of aortic rupture, stroke, spinal chord ischemia, retrograde dissection, endoleaks, aortic dilation > 5mm in diameter

IPD SHARING:
Plan to Share IPD: No
no plan to share data